CLINICAL TRIAL: NCT02916550
Title: Anatomical and Psychophysiological Substrates of Interoception
Brief Title: Breathing Intervention for Cardiac Anxiety
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment rate was lower than anticipated, preventing the study from achieving target sample size.
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Collaborators: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Laureateinstitute
Record Dates: First submitted 2016-09-26; First posted 2016-09-27 (Estimated); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Atrial Fibrillation; Implantable Cardioverter Defibrillator
MeSH Terms: conditions — Atrial Fibrillation | interventions — Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Breathing exercise (Experimental): Participants will perform a paced breathing intervention (slow breathing) prompted by pseudorandomized remote reminders (scheduled reminders plus non scheduled reminders), through cellular phone application.
  Interventions: Behavioral: Breathing exercise

INTERVENTIONS:
Behavioral: Breathing exercise — Participants will perform a paced breathing intervention (slow breathing) prompted by pseudorandomized remote reminders (scheduled reminders plus non scheduled reminders), through cellular phone application.

SUMMARY:
This study examines the impact of a breathing training intervention on cardiorespiratory sensations and anxiety in adults with cardiac arrhythmias.

DETAILED DESCRIPTION:
Patients with cardiac arrhythmias develop increased rates of anxiety and depression. Atrial arrhythmias, such as paroxysmal atrial fibrillation (AF), and ventricular arrhythmias, such as those with implantable cardioverter defibrillators (ICD) are particularly at risk. While ICDs can be life saving, many patients (including those without prior psychiatric illness) develop elevated rates of anxiety and depression, particularly after receiving discharges (shocks) from the device. Treatments involving modulation of the breath have been shown to improve both psychological and cardiac outcomes in patients with AF. Since breathing modulation alters sympathetic balance, this may be a mechanism of the therapeutic effect. This study examines the impact of a breathing training intervention on cardiorespiratory sensations and anxiety in adults with atrial and ventricular cardiac arrhythmias.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80
* BMI 17 to 35
* Proficient in English language
* Paroxysmal atrial fibrillation or ventricular fibrillation or frequent premature atrial/ventricular contractions

Exclusion Criteria:

* No telephone access
* Active suicidal ideation with intent or plan
* Active drug or alcohol dependence, or active binge drinking within the last month
* Cardiovascular instability, as evidenced any of the following:

  1. New York Heart Association (NHYA) heart failure class IV (i.e., unable to carry on any physical activity without discomfort, symptoms of heart failure at rest, increased discomfort with any physical activity is undertaken)
  2. American College of Cardiology/American Heart Association congestive heart failure stage D (i.e., heart failure symptoms at rest, receiving end of life care).
  3. Unstable angina or exercise induced angina
  4. Persistent atrial fibrillation
* Pacemakers or combined pacemaker/ICDs will be excluded
* Presence of unstable cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, or metabolic disease; or any other condition that, in the opinion of the investigator, would make participation not be in the best interest (e.g., compromise the well-being) of the subject or that could prevent, limit, or confound the protocol-specified assessments.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-09; Primary Completion 2021-09 (Actual); Study Completion 2023-05 (Actual)

PRIMARY OUTCOMES:
Cardiac anxiety | 1 month
  Assessed via the Cardiac Anxiety Questionnaire

SECONDARY OUTCOMES:
Disability | 1 month
  Measured by the WHO Disability Assessment Scale (WHODAS)
Wellbeing | 1 month
  NIH Patient Reported Outcome Measurement Information System (PROMIS)
ICD anxiety | 1 month
  Florida Shock Anxiety Scale
Arrhythmia burden | 1 month
  Presence of atrial fibrillation or ICD shocks

CONTACTS AND LOCATIONS:
Overall Officials: Sahib Khalsa, MD, PhD, Principal Investigator — Laureate Institute for Brain Research
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
Not IPD, just de-identified data.